CLINICAL TRIAL: NCT06075004
Title: A Randomized Comparison Between Total Periarticular Anesthetic Infiltration and Partial Posterior Periarticular Anesthetic Infiltration Plus Low Volume Ultrasound-Guided Pericapsular Nerve Group Block for Total Hip Replacement Analgesia
Brief Title: Total Periarticular Infiltration Vs Posterior Periarticular Infiltration Plus PENG Block for Hip Analgesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Daniela Bravo Advis, Principal Investigator, University of Chile
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OAIC 1379/23
Record Dates: First submitted 2023-10-03; First posted 2023-10-10 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Hip Osteoarthritis; Postoperative Pain
Keywords: Nerve block; Periarticular infiltration; Hip replacement; Early rehabilitation
MeSH Terms: conditions — Osteoarthritis, Hip; Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Prospective randomized comparison between two analgesic techniques
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Periarticular Local Anesthetic Infiltration (Active Comparator): 60 mL of 0.25% bupivacaine with 5ug/mL epinephrine will be deposited under direct vision during surgery at the periarticular level before wound closure.
  Interventions: Procedure: Periarticular Local Anesthetic Infiltration
- Posterior Periarticular Local Anesthetic Infiltration plus Pericapsular Nerve Group Block (Experimental): 45 mL of 0.25% bupivacaine with 5ug/mL epinephrine will be deposited under direct vision during surgery at the posterior periarticular level before wound closure.
  After wound closure, an ultrasound-guided pericapsular nerve group block of the hip will be performed using ten mL of 0.5% bupivacaine with 5ug/mL epinephrine.
  Interventions: Procedure: Posterior Periarticular Local Anesthetic Infiltration plus Pericapsular Nerve Group Block

INTERVENTIONS:
Procedure: Periarticular Local Anesthetic Infiltration — Sixty milliliters of 0.25% bupivacaine + 5ug/mL epinephrine and ketorolac 30 mg will be deposited by the orthopedic surgeon at the periarticular level under direct vision during surgery. Fascia, subcutaneous tissues, and skin will also be infiltrated with part of the solution before wound closure.
  Arms: Periarticular Local Anesthetic Infiltration
Procedure: Posterior Periarticular Local Anesthetic Infiltration plus Pericapsular Nerve Group Block — From a total of forty-five milliliters of 0.25% bupivacaine + 5ug/mL epinephrine and ketorolac 30 mg, 15mL will be deposited by the orthopedic surgeon at the posterior periarticular level under direct vision during surgery. Fascia, subcutaneous tissues, and skin will also be infiltrated with part of the solution before wound closure with the remaining 30mL.
  After wound closure, an ultrasound-guided pericapsular nerve group block will be performed by an anesthesiologist by injecting 10mL of 0.5% bupivacaine + 5ug/mL epinephrine in the plane between the iliac bone periosteum and the tendon of the iliopsoas muscle.
  Arms: Posterior Periarticular Local Anesthetic Infiltration plus Pericapsular Nerve Group Block

SUMMARY:
In a recent study, direct periarticular local anesthetic infiltration (PAI) showed a greater incidence of early quadriceps weakness (33% at 3 hours and 13% at 6 hours) than pericapsular nerve group block (PENGB) in total hip arthroplasty (THA) but, in turn, demonstrated a statistically significant better pain control. Additionally, PENGB could not completely circumvent motor compromise either, particularly at 3 hours (20% incidence), probably secondary to an injectate migration towards the femoral nerve. Posteriorly to this publication, a cadaveric trial looking into the maximum effective volume that spared the femoral nerve resulted in 13.2 mL.

This newer evidence led to the design of a strategy that combines both interventions, aiming to obtain the best of them and have a solid alternative for those cases where very early mobilization is pursued.

Thus, it is hypothesized that posterior PAI added to a low-volume PENGB (10mL) represents a superior alternative to PAI in terms of strength preservation and provides effective analgesia during the first 24 postoperative hours after THA.

DETAILED DESCRIPTION:
Patients who agree to participate in the protocol will be assigned to one group or another (PAI or posterior PAI+PENGB) through computationally generated block randomization. Outcome assessors blinded to randomization will perform all measurements.

All trial interventions (PAI or posterior PAI+PENGB) will be performed (or supervised) by one of the co-authors, an expert orthopedic surgeon anesthesiologist. Both interventions will be executed in the operating room, on the surgical table, under sedation, and with the barrier that separates the surgical field from the cranial area of the patient to keep the latter blind to the technique received.

All patients will undergo spinal anesthesia using 0.5% bupivacaine (10mg) plus 20 μg of fentanyl. Both groups will also receive tranexamic acid 1g intravenous (IV), ketoprofen 100mg IV, and acetaminophen 1gr IV. Propofol sedation guided with a targeted controlled infusion (TCI) model will be administered in order to obtain an adequate level of sedation.

All surgeries will be conducted by the same team of surgeons, performing a posterior approach technique in the lateral decubitus position.

In the recovery room, all patients will receive patient-controlled analgesia (morphine bolus = 1 mg; lockout interval = 8 minutes). On the surgical ward, all subjects will continue to receive acetaminophen (1 g per os every 6 hours), ketoprofen (100 mg per os every 8 hours) as well and patient-controlled analgesia (morphine bolus = 1 mg IV; lockout interval = 8 minutes).

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists classification 1-3
* Body mass index between 20 and 35 (kg/m2)

Exclusion Criteria:

* Adults who are unable to give their own consent
* Pre-existing neuropathy (assessed by history and physical examination)
* Coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work-up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or prothrombin time ≥ 50)
* Renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work-up i.e. creatinine ≥ 100)
* Hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work-up i.e. transaminases ≥ 100)
* Allergy to local anesthetics (LAs) or morphine
* Pregnancy
* Prior surgery in the inguinal area corresponding surgical side
* Chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-10-23 (Estimated)

PRIMARY OUTCOMES:
Presence of quadriceps motor block (defined as paralysis or paresis) | 3 hours after post anesthesia care unit (PACU) arrival
  Quadriceps motor function will be tested with the patient lying on the bed and with the hip joint at 45º and the knee at 90º. The subject will be asked to extend the knee, first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).

SECONDARY OUTCOMES:
Presence of quadriceps motor block (defined as paralysis or paresis) | 6 hours after post anesthesia care unit (PACU) arrival
  Quadriceps motor function will be tested with the patient lying on the bed and with the hip joint at 45º and the knee at 90º. The subject will be asked to extend the knee, first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Presence of quadriceps motor block (defined as paralysis or paresis) | 24 hours after post anesthesia care unit (PACU) arrival
  Quadriceps motor function will be tested with the patient lying on the bed and with the hip joint at 45º and the knee at 90º. The subject will be asked to extend the knee, first against gravity and then against resistance. Quadriceps strength will be graded according to a 3-point scale: normal strength = 0 point (extension against resistance); paresis = 1 point (extension against gravity but not against resistance); and paralysis = 2 points (no extension).
Hip adduction strength | 3 hours after post anesthesia care unit (PACU) arrival
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1, and 2 points as decreases in strength of 0-20% (normal strength), 21-70% (paresis), and 71-90% (paralysis) compared to the baseline measurement, respectively.
Hip adduction strength | 6 hours after post anesthesia care unit (PACU) arrival
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1, and 2 points as decreases in strength of 0-20% (normal strength), 21-70% (paresis), and 71-90% (paralysis) compared to the baseline measurement, respectively.
Hip adduction strength | 24 hours after post anesthesia care unit (PACU) arrival
  Hip adduction will be evaluated by comparing it to baseline strength (i.e., prior to spinal anesthesia). A blood pressure cuff, inflated at 40 mmHg, will be inserted between the knees of the patient: the latter will then be instructed to squeeze the cuff as hard as possible and to sustain the effort. We will define hip adduction scores of 0, 1, and 2 points as decreases in strength of 0-20% (normal strength), 21-70% (paresis), and 71-90% (paralysis) compared to the baseline measurement, respectively.
Postoperative morphine consumption | 24 hours after PACU arrival
  Consumption of intravenous morphine (mg) registered by a patient-controlled analgesia device.
Postoperative morphine consumption | 48 hours after PACU arrival
  Consumption of intravenous morphine (mg) registered by a patient-controlled analgesia device.
Time until first morphine demand | 48 hours after PACU arrival
  Time (minutes) until first patient-controlled analgesia morphine demand.
Static and dynamic pain | 3 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain).
Static and dynamic pain | 6 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain).
Static and dynamic pain | 12 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain).
Static and dynamic pain | 18 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain).
Static and dynamic pain | 24 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain).
Static and dynamic pain | 48 hours after PACU arrival
  Pain intensity at rest and during active movement (hip adduction) using a numeric rating score (NRS) ranged from 0 to 10 (0 = no pain and 10 = worst imaginable pain).
Sensory block | 3 hours after PACU arrival
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch).
Sensory block | 6 hours after PACU arrival
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch).
Sensory block | 24 hours after PACU arrival
  Sensory block in the anterior, lateral and medial aspects of the mid-thigh. For each territory, blockade will be evaluated using a 3-point scale: 0 = no block, 1 = analgesia (patient can feel touch, not cold), 2 = anesthesia (patient cannot feel touch).
Block/Infiltration-related complications | 1 hour after nerve block or local anesthetic infiltration
  Incidence of adverse events related to nerve block or local anesthetic infiltration (i.e. vascular puncture, local anesthetic systemic toxicity).
Postoperative opioid related side effects | 48 hours after PACU arrival
  Presence of postoperative nausea, vomiting, pruritus, urinary retention, respiratory depression.
Duration of surgery | 4 hours after skin incision
  Time between skin incision and closure (min).
Inability to perform physiotherapy due to motor block | 6 hours after PACU arrival
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to decreased strength in the operated limb.
Inability to perform physiotherapy due to motor block | Postoperative day 1
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to decreased strength in the operated limb.
Inability to perform physiotherapy due to motor block | Postoperative day 2
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to decreased strength in the operated limb.
Inability to perform physiotherapy due to pain | 6 hours after PACU arrival
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to pain in the operated limb.
Inability to perform physiotherapy due to pain | Postoperative day 1
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to pain in the operated limb.
Inability to perform physiotherapy due to pain | Postoperative day 2
  Number of participants that cannot end the physiotherapy protocol programmed for the sixth hour after PACU arrival secondary to pain in the operated limb.
Readiness to discharge | 4 days after surgery
  Days to be ready for discharge following physiotherapist criteria
Length of hospital stay | 7 days after surgery
  Length of hospital stay after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Bravo, MD, Principal Investigator — University of Chile
Locations (1):
- Hospital Clínico Universidad de Chile, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Wainwright TW, Gill M, McDonald DA, Middleton RG, Reed M, Sahota O, Yates P, Ljungqvist O. Consensus statement for perioperative care in total hip replacement and total knee replacement surgery: Enhanced Recovery After Surgery (ERAS(R)) Society recommendations. Acta Orthop. 2020 Feb;91(1):3-19. doi: 10.1080/17453674.2019.1683790. Epub 2019 Oct 30. PMID 31663402
- [Background] Giron-Arango L, Peng PWH, Chin KJ, Brull R, Perlas A. Pericapsular Nerve Group (PENG) Block for Hip Fracture. Reg Anesth Pain Med. 2018 Nov;43(8):859-863. doi: 10.1097/AAP.0000000000000847. PMID 30063657
- [Background] Kuchalik J, Magnuson A, Lundin A, Gupta A. Local infiltration analgesia or femoral nerve block for postoperative pain management in patients undergoing total hip arthroplasty. A randomized, double-blind study. Scand J Pain. 2017 Jul;16:223-230. doi: 10.1016/j.sjpain.2017.05.002. Epub 2017 Jun 1. PMID 28850408
- [Background] Bravo D, Aliste J, Layera S, Fernandez D, Erpel H, Aguilera G, Arancibia H, Barrientos C, Wulf R, Leon S, Branes J, Finlayson RJ, Tran Q. Randomized clinical trial comparing pericapsular nerve group (PENG) block and periarticular local anesthetic infiltration for total hip arthroplasty. Reg Anesth Pain Med. 2023 Oct;48(10):520-521. doi: 10.1136/rapm-2023-104487. Epub 2023 Mar 22. No abstract available. PMID 36948525
- [Background] Leurcharusmee P, Kantakam P, Intasuwan P, Malatong Y, Maikong N, Navic P, Kitcharanant N, Mahakkanukrauh P, Tran Q. Cadaveric study investigating the femoral nerve-sparing volume for pericapsular nerve group (PENG) block. Reg Anesth Pain Med. 2023 Nov;48(11):549-552. doi: 10.1136/rapm-2023-104419. Epub 2023 Apr 7. PMID 37028817